CLINICAL TRIAL: NCT06340022
Title: Comparison of Pain and Anxiety Levels of Sleeperone 5 Electronic Anesthesia System and Conventional Local Anesthesia Techniques in Pediatric Patients: a Randomised Clinical Study
Brief Title: Pain and Anxiety Levels of Sleeperone Electronic Anesthesia System in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Irem Bag, Assoc.Prof., Eskisehir Osmangazi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2022-31
Record Dates: First submitted 2024-03-18; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Dental Anxiety; Pain
Keywords: Dental Anxiety; Intraosseous Anesthesia; Pain; SleeperOne
MeSH Terms: conditions — Pain | interventions — Weights and Measures; Heart Rate

STUDY DESIGN:
Intervention Model Description: The study was a single-center randomized controlled trial using a split mouth design with a 1:1 split ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upper jaw (Experimental): * A half of upper jaw: Electronic local anesthesia technique (SleeperOne) A topical anesthetic spray containing 10% lidocaine was applied with a cotton pellet for 1 minute.The SleeperOne® 5 (Dentalhitec, Mazières-en-Mauges, France) device was used with 30 gauge-0.30x09 mm Effitec needle tips for intraosseous anesthesia. The anesthesia was applied in child mode according to the manufacturer.1 ml of local anesthetic solution (Ultracaine D-S Fort) was applied for 1 minute.
  * The contralateral half of the upper jaw: Infiltrative anesthesia (conventional) After confirming the vitality of the tooth, a topical anesthetic spray was applied with a cotton pellet for 1 minute. A local anesthetic, Maxicaine Forte, was administered for 1.5 ml for 1 minute using buccal infiltration anesthesia technique using short syringes.
  Interventions: Other: Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) scale; Other: Face Image Scale (FIS) scoring system; Other: Visual Analogue Scale (VAS); Other: pulse rate
- Lower jaw (Experimental): * A half of lower jaw: Electronic local anesthesia technique (SleeperOne) A topical anesthetic spray containing 10% lidocaine was applied with a cotton pellet for 1 minute.The SleeperOne® 5 (Dentalhitec, Mazières-en-Mauges, France) device was used with 30 gauge-0.30x09 mm Effitec needle tips for intraosseous anesthesia. The anesthesia was applied in child mode according to the manufacturer.1 ml of local anesthetic solution (Ultracaine D-S Fort) was applied for 1 minute.
  * The contralateral half of the lower jaw: mandibular anesthesia (conventional) After topical anesthesia, mandibular anesthesia with Maxicaine Forte,in an amount of 1.8 ml was administered for 1 minute using long syringes.
  Interventions: Other: Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) scale; Other: Face Image Scale (FIS) scoring system; Other: Visual Analogue Scale (VAS); Other: pulse rate

INTERVENTIONS:
Other: Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) scale — Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) scale was applied to determine the anxiety level before the procedure.
Other: Face Image Scale (FIS) scoring system — Face Image Scale (FIS) scoring system (1= not afraid at all, 2= very little afraid, 3= afraid, 4= quite afraid, 5= very much afraid) was used to determine the anxiety level before starting anesthesia and after the anesthesia.
Other: Visual Analogue Scale (VAS) — In the Visual Analogue Scale (VAS), the patient was asked to rate the pain he/she felt during anesthesia on a 10 cm long ruler ranging from no pain=0 to unbearable pain=10.
Other: pulse rate — Before starting anesthesia and after the anesthesia the patient's pulse rate was measured and recorded with a pulse oximeter.

SUMMARY:
The conventional method used for dental anesthesia in children is the administration of a local anesthetic solution by injection. Although this process successfully eliminates pain during the procedure, it continues to be a problem for many children in terms of dental anxiety before and during anesthesia administration.

The aim of this study is to compare intraosseous anesthesia with SleeperOne® 5, a computer-assisted local anesthesia system, with conventional local anesthesia techniques in terms of pain and anxiety.

DETAILED DESCRIPTION:
In the conventional injection technique, painful local swelling of the tissues at the injection site occurs during the administration of local anesthetics. Failure to control the rate of administration of anesthesia increases pain, swelling and tissue tension, leading to the discomfort and unpleasant sensations that accompany local anesthesia. In addition, an uncontrolled and shocking increase in pressure in the anesthetized tissues can lead to short-term blood supply disturbances and local damage, reducing the effectiveness of anesthesia and increasing the risk of side effects. It has been reported that the pain felt during anesthesia is mostly caused by the inability to control the pressure generated during the injection of the solution. To overcome these shortcomings, the search for new alternative and minimally invasive methods of local anesthesia has been in the limelight with better pain control, reduced injection pain and improved quality of treatment for pedodontic procedures. With the use of computer-assisted local anesthesia systems, the anesthetic solution is administered gradually and the tissue pressure during anesthesia can be controlled. Thus, a less painful and more comfortable anesthesia experience can be provided. SleeperOne® 5, one of the computer-assisted local anesthesia systems, is a device with advantages such as ease of use, less intimidating physical appearance of the needle, no need for pressure during injection, guided entry points to the injection site. There are no previous studies comparing the use of intraosseous technique with SleeperOne® 5 device and conventional mandibular anesthesia in mandibular permanent molars. In this study, the investigators aimed to compare the pain and anxiety caused by the SleeperOne® 5 anesthesia system in children compared to traditional anesthesia methods, of which there are few studies in the literature. The first null hypothesis (H0) of the study is that there is no difference between intraosseous anesthesia administered with SleeperOne® 5 computer-assisted anesthesia systems and buccal infiltration and mandibular anesthesia administered with conventional methods in terms of anxiety in patients. The second null hypothesis of the study is that there is no difference between intraosseous anesthesia performed with SleeperOne® 5 computer-assisted anesthesia systems and buccal infiltration and mandibular anesthesia performed with conventional methods in terms of pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA 1 general systemic status
* Patients aged 8-12 years
* Patients in Frankl behavior rating score of III and IV
* Asymptomatic teeth
* Patients with carious lesions not exceeding 1/3 of the buccolingual distance between the buccal and lingual pulp crests on the occlusal surfaces of right and left upper/lower permanent first molars with complete apical root development
* Patients with permanent first molars with caries at a minimum dentin 1/2 level and intact dentin at the pulp margin on radiographic evaluation

Exclusion Criteria:

* Patients with mild or severe systemic disease, receiving medical treatment
* Patients younger than 8 years and older than 12 years
* Uncooperative, non-compliant patients in the Class I or Class II group according to the Frankl behavior scale
* Teeth with a history of spontaneous pain and tenderness on palpation and percussion
* Patients in need of dental treatment requiring urgent intervention
* Teeth with incomplete apical root development
* Patients with large carious lesions that exceed 1/3 of the distance between the occlusal and buccolingual pulp crests
* Patients with teeth with clinical or radiographic evidence of caries on the interdental or buccal and/or lingual surfaces
* Teeth with caries lesions that do not reach dentin 1/2 on radiographic evaluation or teeth with intact dentin tissue at the pulpal margin

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
The pulse rate measurements before and after the anesthesia techniques | 7 months
  Application and recording of scale measurements of pulse rate before and after the anesthesia techniques (normal 70-120 bpm)
Determine the anxiety level before the procedures | 7 months
  Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) scale before the anesthesia procedures. A score between 1 and 5 was made according to the answers given to each question in this scale (1 point = not at all afraid, 2 points = slightly afraid, 3 points = moderately afraid, 4 points = quite afraid, 5 points = very afraid). If the score obtained from the CFSS-DS measurement results is below 38, it is considered as non-anxious, between 38-45 as significant dental anxiety, and as 45 and above as high level dental anxiety.
The anxiety measurements before and after the anesthesia techniques | 7 months
  Application and recording of scale measurements of Face Image Scale (FIS) scoring system before and after the anesthesia techniques.(1= not afraid at all, 2= very little afraid, 3= afraid, 4= quite afraid, 5= very much afraid)
The pain measurements during the anesthesia techniques | 7 months
  In the Visual Analogue Scale (VAS), the patient was asked to rate the pain he/she felt during anesthesia on a 10 cm long ruler ranging from no pain=0 to unbearable pain=10. The results were recorded on the forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University Faculty of Dentistry, Department of Pediatric Dentistry, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Other researchers will be able to access the individual participant data from the corresponding author.

REFERENCES:
- [Background] Sixou JL, Marie-Cousin A, Huet A, Hingant B, Robert JC. Pain assessment by children and adolescents during intraosseous anaesthesia using a computerized system (QuickSleeper). Int J Paediatr Dent. 2009 Sep;19(5):360-6. doi: 10.1111/j.1365-263X.2009.00983.x. Epub 2009 Apr 14. PMID 19486372
- [Background] Sovatdy S, Vorakulpipat C, Kiattavorncharoen S, Saengsirinavin C, Wongsirichat N. Inferior alveolar nerve block by intraosseous injection with Quicksleeper(R) at the retromolar area in mandibular third molar surgery. J Dent Anesth Pain Med. 2018 Dec;18(6):339-347. doi: 10.17245/jdapm.2018.18.6.339. Epub 2018 Dec 28. PMID 30637344
- [Background] Beneito-Brotons R, Penarrocha-Oltra D, Ata-Ali J, Penarrocha M. Intraosseous anesthesia with solution injection controlled by a computerized system versus conventional oral anesthesia: a preliminary study. Med Oral Patol Oral Cir Bucal. 2012 May 1;17(3):e426-9. doi: 10.4317/medoral.17543. PMID 22143722
- [Background] Dempsy Chengappa MM, Prashanth AK. Evaluation of efficacy of computer-controlled local anaesthetic delivery system vs traditional injection system for minor pediatric surgical procedures in children. Med J Armed Forces India. 2022 Sep;78(Suppl 1):S89-S95. doi: 10.1016/j.mjafi.2020.08.010. Epub 2020 Nov 2. PMID 36147427
- [Background] Angelo Z, Polyvios C. Alternative practices of achieving anaesthesia for dental procedures: a review. J Dent Anesth Pain Med. 2018 Apr;18(2):79-88. doi: 10.17245/jdapm.2018.18.2.79. Epub 2018 Apr 27. PMID 29744382
- [Background] Versloot J, Veerkamp JS, Hoogstraten J. Computerized anesthesia delivery system vs. traditional syringe: comparing pain and pain-related behavior in children. Eur J Oral Sci. 2005 Dec;113(6):488-93. doi: 10.1111/j.1600-0722.2005.00252.x. PMID 16324138
- [Background] Anil O, Keskin G. Comparison of computer controlled local anesthetic delivery and traditional injection regarding disruptive behaviour, pain, anxiety and biochemical parameters: a randomized controlled trial. J Clin Pediatr Dent. 2024 Jan;48(1):120-127. doi: 10.22514/jocpd.2023.046. Epub 2024 Jan 3. PMID 38239164